CLINICAL TRIAL: NCT06337539
Title: Precision Psychiatry for Depression: Immune Response and Affective Symptoms as Predictors of Response to Antidepressants
Acronym: LYMPHODEP
Status: Not yet recruiting | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PI-23-185
Record Dates: First submitted 2024-02-27; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Depression; Inflammation; Antidepressants; Immunity
Keywords: Selective serotonin reuptake inhibitors; Depression; Inflammation; Immunity
MeSH Terms: conditions — Depression; Inflammation | interventions — Sertraline; Citalopram; Escitalopram; Fluoxetine; Paroxetine; Fluvoxamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Immunological and biochemical variables:
  * Acute phase biomarkers: CRP
  * Proinflammatory cytokines: IL-1, IL-6, TNF-α, IL-12, IL-23, IL-17, IL-22
  * Anti-inflammatory cytokines: IL-10, IL-4, tumor growth factor (TGF) -β
  * Cortisol
  * Oxidative and nitrosative stress: Zinc, Glutathione, Albumin, Uric Acid, Bilirubin, Vitamin C and Vitamin E
  * Microglia activation: microRNA (miR)-155, miR-126, miR-223, miR-146a, miR-21, miR-124
  * Neurogenesis and neuroinflammation: BDNF, VILIP-1, CC chemokine ligand 2 (MCP-1), sTREM-2, vascular endothelial growth factor (VEGF), sTREM-1, β-NGF, sRAGE, CX3CL1
  * Lymphocyte subpopulations in peripheral blood (Th1, Th2, Th17, Th1/17, Treg, naive cells, total Tfh, Tγδ1, Tγδ2, Tγδ17, Tγδ1/17, monocytes)
  * Transcriptomic and proteomic lymphocyte study at the single-cell level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SSRI treatment: The subjects who will participate in this study will be outpatients seen in the Psychiatry Outpatient Clinics of the Germans Trias i Pujol University Hospital (Badalona, Spain) clinically diagnosed with major depression and eligible to receive antidepressant treatment with SSRIs.
  The control group will be made up of healthy subjects, using the same inclusion and exclusion criteria except for the psychiatric diagnosis.
  Interventions: Drug: SSRI

INTERVENTIONS:
Drug: SSRI — Outpatients with a diagnosis of major depression in the Psychiatry Outpatient Clinics will be evaluated for recruitment.
  * Recruitment visit: It will be carried out by one of the psychiatrists participating in the study. The patient will be informed about the study and written consent will be requested. Subsequently, the inclusion and exclusion criteria will be reviewed, and all demographic and clinical variables will be collected.
  * Baseline visit: One of the psychiatrists will interview the patient and apply the semi-structured clinical interview and the psychopathological evaluation questionnaires. In addition, a blood draw will be performed for serum collection, spectral cytometric analysis of lymphocyte subpopulations and obtaining peripheral blood mononuclear cells (PBMCs).
  * Follow-up visit after 3 months of treatment: Clinical variables will be collected and the same procedures will be performed as during the baseline visit. Not in the control group.
  Other Names: Sertraline; Citalopram; Escitalopram; Fluoxetine; Paroxetine; Fluvoxamine

SUMMARY:
Objectives: To identify in patients with major depression different peripheral markers of neuroinflammation in relation to affective symptoms (anxiety, depression, irritability), fatigue and cognitive symptoms; and its relationship with the response to antidepressant treatment with selective serotonin reuptake inhibitors (SSRIs).

Methodology: This is a prospective observational cohort study in patients with major depression naturally subjected to treatment with SSRIs. For this, 30 patients with major depression attended in the Outpatient Psychiatry Consultations will be selected. All of them will be evaluated at baseline and after 3 months of treatment, collecting demographic and clinical variables, Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) psychiatric diagnoses, psychopathological scales and immunological and biochemical variables. The correlation between immunological markers and affective and cognitive symptoms at baseline, as well as their variation with treatment, will be analyzed. A group of 20 healthy subjects will be used as a control group.

Subsequently, a bivariate comparative analysis will be carried out, where the statistically significant or marginally significant variables associated with psychopathological variables will be used to build a multivariate binary logistic regression model.

DETAILED DESCRIPTION:
Depression is the mental disorder that has the highest prevalence, affecting approximately 16% of the general population and having a great impact on the global functionality of patients. According to the World Health Organization (WHO), depression will be considered the main cause of disability in 2030. At the end of the last century, a large part of the studies on the neurobiological bases of depression evolved from the monoaminergic hypothesis. This theory proposes that the etiopathogenesis of depression would be directly related to a reduction in monoaminergic activity (noradrenergic, serotonergic or both) in the central nervous system (CNS). From there, it was postulated that the antidepressant action of various drugs could be due to an enhancement of neurotransmission as a consequence of the increase in the concentration of monoamines at the level of the synaptic space. This monoaminergic hypothesis, however, does not answer some important questions such as what causes these monoaminergic alterations? Or how do we explain the existence of 30% of patients refractory to antidepressant treatment? For this reason, there has been growing interest in recent years in other theories that focus on the immune and endocrine systems.

The immune system and the nervous system share the functions of recognizing objects, discerning their qualities and generating an adaptive response related to them. The inflammatory reflex (innate immunity) depends on the detection of specific molecular patterns in invaders, but not expressed by own tissues. One of the first observations on the relationship of the innate immune system to the CNS was the increase in blood concentrations of inflammatory biological markers, such as C-reactive protein (CRP) and fibrinogen, in patients with depression. Since then, and especially in the field of major depression, there is a growing body of literature supporting its link with inflammation: frequent comorbidity with inflammatory diseases such as coronary heart disease or rheumatoid arthritis; presence of elevated levels of proinflammatory cytokines; potential of exogenous proinflammatory cytokines to induce depressive symptoms; the association of levels of peripheral markers of inflammation with the severity of depression; potential of antidepressants to inhibit inflammation; antidepressant effects of anti-inflammatory agents such as nonsteroidal anti-inflammatory drugs (NSAIDs), etc. In addition to proinflammatory molecules, alterations in the levels of lymphocyte subpopulations such as T helper type 17 (Th17) or T regulatory cells (Treg) have recently been characterized in patients with major depression that could be related to the neuroinflammatory process.

The impact of inflammation on behavior, however, is not only associated with depression itself, but with specific dimensions of symptoms such as alterations in motivation and motor activity (fatigue, psychomotor impairment) and with greater sensitivity to the threat (anxiety, arousal, alarm).

The results of this project will contribute, first of all, to a better understanding of the immunological aspects of depressive processes, which will favor the possibility of developing new targets for future treatments of this disease. Secondly, the results will help identify biological and clinical markers that predict response to antidepressant treatment.

Hypothesis

1. The combination of immune response biomarkers (acute phase inflammation, cytokines, hypothalamic-pituitary-adrenal (HPA) axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes, Treg and neurogenesis), symptoms of positive and negative valence systems of Research Domain Criteria (RDoC) (depression, anhedonia, fatigue, anxiety) and cognitive dysfunction allows to establish a prediction about the response to treatment with SSRI antidepressants in patients with major depression.
2. Symptoms included in RDoC positive and negative valence systems (depression, anhedonia, fatigue, anxiety), as well as cognitive dysfunction, are positively related to biomarkers of acute phase inflammation, proinflammatory cytokines, HPA axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes and negatively related to biomarkers of anti-inflammatory cytokines, Treg and neurogenesis in patients with major depression compared to healthy controls.
3. The improvement of symptoms included in the positive and negative valence systems of RDoC (depression, anhedonia, fatigue, anxiety) as well as cognitive dysfunction after antidepressant treatment with SSRIs are related to the reduction of biomarkers of acute phase inflammation, proinflammatory cytokines, HPA axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes, and increased anti-inflammatory cytokines, Treg and neurogenesis.

Primary Objective

1. To assess the combination of immune response biomarkers (acute phase inflammation, cytokines, HPA axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes, Treg and neurogenesis), symptoms of positive and negative valence systems of RDoC (depression, anhedonia, fatigue, anxiety) and cognitive dysfunction as predictors of response to SSRI antidepressant treatment in patients with major depression.

   Secondary Objectives
2. To evaluate the relationship between biomarkers of immune response (acute phase inflammation, cytokines, HPA axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes, Treg and neurogenesis) and symptoms of the positive and negative valence systems of RDoC (depression, anhedonia, fatigue, anxiety) and cognitive dysfunction in patients with major depression compared to healthy controls.
3. To evaluate the relationship between biomarkers of immune response (acute phase inflammation, cytokines, HPA axis, oxidative and nitrosative stress, activation of microglia and Th17 and Tγδ17 lymphocytes, Treg and neurogenesis) and symptoms of the positive and negative valence systems of RDoC (depression, anhedonia, fatigue, anxiety) and cognitive dysfunction in patients with major depression in relation to response to treatment.
4. To define the phenotype and transcriptome of the lymphocyte subpopulations of patients with major depression before and after treatment.
5. To evaluate the kinetics of the lymphocyte subpopulations of patients with major depression at different times of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Clinical diagnosis of major depression according to DSM-5 criteria made by a psychiatrist applying the Structured Clinical Interview for DSM-5 (SCID-5).
* Eligible for receiving antidepressant treatment for major depression.

Exclusion Criteria:

* Who have received antidepressant, antipsychotic or euthymizer treatments in the 6 weeks prior to inclusion in the study.
* Who present concurrent psychotic symptoms.
* Who present disorders due to alcohol or drug use, with active consumption during the last 3 months.
* Pregnant women.
* Who have serious or unstable medical disorders, Addison's or Cushing's disease, systemic inflammatory or autoimmune diseases, or primary or secondary immunodeficiencies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects that will participate in this study will be outpatients attended in the Outpatient Psychiatry Consultations of the Hospital Universitari Germans Trias i Pujol (Badalona, Spain) clinically diagnosed with major depression and eligible to receive antidepressant treatment with SSRIs. The control group will be made up of healthy subjects, using the same inclusion and exclusion criteria except for the psychiatric diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Response | 3 months
  The response to treatment will be assessed using the Montgomery-Åsberg Depression Rating Scale (MADRS) scale scores. The MADRS scoring instructions indicate that a total score ranging from 0 to 6 indicates that the patient is in the normal range (no depression), a score ranging from 7 to 19 indicates "mild depression", 20 to 34 indicates "moderate depression", a score of 35 and greater indicates "severe depression", and a total score of 60 or greater indicates "very severe depression".

SECONDARY OUTCOMES:
Lymphocyte subpopulations | 3 years
  For the study of lymphocyte subpopulations, a multidimensional flow cytometry panel has been designed. The panel includes markers for the identification of the most representative subpopulations of T cells (Th1, Th2, Th17, Th1/17, Treg, naïve cells, central memory and effector memory, total Tfh, Tγδ1, Tγδ2, Tγδ17, Tγδ1/17...) and monocytes as well as activation markers (HLADR, CD38), inhibitory checkpoints (PD1, TIM3) and markers of tissue migration and response to chemokines (CCR2, CX3CR1, CXCR6). The results of expression markers and subpopulations will be expressed as percentage over total lymphocyte counts.
Biochemical variables | 3 years
  From the serum samples, the analysis of C-reactive protein and immunoglobulins will be performed by Chemiluminescence immunoassay and expressed in mg/dl. The study of pro-inflammatory and anti-inflammatory cytokines (IL-1, IL-6, Tumor Necrosis Factor (TNF)-α, Interleukin (IL)-12, IL-23, IL-17, IL-22, TGFbeta, IL-10, IL-4) and neurogenesis/neuroinflammation factors (BDNF, VILIP-1, β-Nerve Growth Factor (NGF), sRAGE, chemokine C-X3-C motif ligand 1 (CX3CL1), Soluble triggering receptor expressed on myeloid cell-2 (sTREM-2)) in serum using Multiplex Bead-based Immunoassay technology and expressed in pg/ml. The study of the relative expression of miRNAs (miR-155, miR-126, miR-223, miR-146a, miR-21, miR-124) will also be carried out from serum samples using real time quantitative PCR (RT-qPCR).
Single-cell CITEseq | 3 years
  Frozen samples will be used to perform lymphocyte transcriptomic and proteomic study at the single cell level, allowing the study of the immune system in great depth. For this, Single cell RNA sequencing technology (CITEseq) will be used. CITEseq is a multimodal single-cell phenotyping method that uses antibody-bound oligonucleotides that act as synthetic transcripts that are captured during single-cell RNA-seq library preparation protocols. This allows immunophenotyping of cells with a potentially unlimited number of markers and analysis of the transcriptome using single-cell sequencing approaches such as those developed by 10x Genomics.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Iglesias-González, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided